CLINICAL TRIAL: NCT04501887
Title: The Efficacy of Precision Treatment for Gastric Cancer Guided by Multidimensional Molecular Biology Profiling: a Multi-center Clinical Study
Brief Title: The Efficacy of Precision Treatment for Gastric Cancer Guided by Molecular Profiling
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Tianshu Liu, Doctor, Shanghai Zhongshan Hospital
Other Study IDs: ZS-ON-100
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; precision medicine
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Matched therapy: Molecular profiling performed with actionable molecular alterations detected and target therapy was then conducted
- Unmatched therapy: Molecular profiling performed with actionable molecular alterations detected but therapy was conducted based on the guideline treatment
- No marker: Molecular profiling performed without any actionable molecular alterations detected, tranditional therapy based on the guideline was then conducted

SUMMARY:
Gastric cancer (GC) is one of the most common and lethal cancers worldwide, especially in China, and the median overall survival for patients with advanced, metastatic GC remains only about 1 year. Several molecular profiling studies have demonstrated that a proportion of gastric cancer harbour actionable molecular alterations which shows a predictive benefit from a specific therapy (in any cancer type). In the current study, the efficacy of precision treatment for gastric cancer guided by multidimensional molecular biology profiling will be observed. The analysis focused on the overall survival outcomes for patients whose tumours harboured actionable molecular alterations and who received appropriately matched therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female. Age: 18-80 years.
2. Histologically confirmed adenocarcinoma of the stomach or gastro-esophageal junction with inoperable locally advanced or recurrent and/or metastatic disease, not amenable to curative therapy.
3. Measurable disease, according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, assessed using imaging techniques (CT or MRI).
4. Multidimensional molecular biology profiling has been conducted using tumor or blood sample.
5. ECOG Performance status 0-1.
6. Life expectancy of at least 3 months.
7. Signed informed consent.

Exclusion Criteria:

1. The quality of NGS reports does not fit the requirement.
2. History of documented congestive heart failure; angina pectoris requiring medication; evidence of transmural myocardial infarction on ECG; poorly controlled hypertension (systolic BP > 180 mmHg or diastolic BP > 100 mmHg); clinically significant valvular heart disease; or high risk uncontrollable arrhythmias.
3. Baseline LVEF < 50% (measured by echocardiography or MUGA).
4. Patients with dyspnea at rest due to complications of advanced malignancy or other disease, or who require supportive oxygen therapy.
5. Patients receiving chronic or high dose corticosteroid therapy. (Inhaled steroids and short courses of oral steroids for anti-emesis or as an appetite stimulant are allowed).
6. Known dihydropyrimidine dehydrogenase (DPD) deficiency.
7. History or clinical evidence of brain metastases.
8. Serious uncontrolled systemic intercurrent illness, e.g. infections or poorly controlled diabetes.
9. Positive serum pregnancy test in women of childbearing potential.
10. Subjects with reproductive potential not willing to use an effective method of contraception.
11. Major surgery within 4 weeks of start of study treatment, without complete recovery.
12. Patients with known active infection with HIV, HBV, or HCV.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy-confirmed gastric cancer at stage IV who conducted molecular testing are included.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | up to 3 years
  Overall survival was measured from the date of advanced disease until death.
Progression-free survival | up to 3 years
  The PFS was calculated from the date of advanced disease to the date of disease progression or death

SECONDARY OUTCOMES:
Positive rate | up to 3 years
  Actionable molecular alterations detected by molecular profiling